CLINICAL TRIAL: NCT06065644
Title: Inducible Displacements of the Sacroiliac Joint Measured With CTMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bergen (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IDSCT
Record Dates: First submitted 2022-11-03; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Sacroiliac Joint Unstable
Keywords: CT method; low dose CT; Sacroiliac joint; CT-RSA; CTMA; IMA

STUDY DESIGN:
Intervention Model Description: 15 patients with long fixation and 15 with fixation of L4/5.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long fixation (Experimental): CT in a neutral and then by provocation (anterior straight leg raise and figure-of-four).
  Interventions: Device: CTMA
- One segment fixation (Active Comparator): CT in a neutral and then by provocation (anterior straight leg raise and figure-of-four).
  Interventions: Device: CTMA

INTERVENTIONS:
Device: CTMA — Induced displacement of the Sacroiliac joint

SUMMARY:
To evaluate the influence of different surgical treatment options for kyphoscoliosis we measure the movement of the SI joint with Radiostereometric analysis (RSA) after lumbar fixation with CT motion analysis (CTMA).

DETAILED DESCRIPTION:
CTMA is a high precision in vivo measuring method for motion. We intend to measure sacroiliac joint (SIJ) movement in long fixations compared to short fixations. The Center for Implant and Radiostereometric Research Oslo (CIRRO) has extensive experience with RSA and established state of the art measuring method of movement in the SIJ. We have compared the methode with CTMA and established a methode for CTMA measurements at CIRRO. We will measure the movement in the SIJ in patients that have long fixations of 3 or more segments down to S1 and compare it to one segment fixation in the level of L4/5. Null hypothesis

* The SI movement will not increase because of long fixation down to sacrum, the SIJ will not work as an adjacent level and not compensatory increase the movement.
* The increased movement will not result in low back pain and /or pseudo radicular pain to the lower limbs CTMA is a high accuracy measuring method comparable to RSA. With a precision of RSA of 1 degree for rotation we need 10 patients in each group to detect a difference of 2 degrees for power of 90% on an alpha = 99% confidence level. Taking drop-outs into account we need a group size of 15 resulting in 30 patients (Two- sided T-test).

ELIGIBILITY:
Inclusion Criteria:

* Long fixations of 3 or more segments down to S1, (also including not correction surgery patients).
* One segment fixations in the level of L4/5 regardless of olisthesis.

Exclusion Criteria:

* Medical conditions that affect the SI joint (Sacroileitis, Ankylosing spondylitis, psoriasis, autoimmune illness)
* Do not want to participate and not able to answer PROMs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Movement | 12 months
  Compare the induced movement of the SIJ joint Movement measured in millimeter around x, y, z axis 3 dimensional and usually in the range of -2-2 millimeters when comparing neutral position to provoked position.

SECONDARY OUTCOMES:
Oswestry disability index | 12 months
  From the Norwegian quality register for spinal surgery. 0-20% minimal disability, 21-40% moderate disability, 41-60% sever disability, 61-80% crippled, 81-100% bed bound
EQ 5D 5L | 12 months
  From the Norwegian quality register for spinal surgery. EQ-5D health states; When a person completes the EQ-5D questionnaire, the descriptive system produces a 5-digit health status profile that represents that person's level of reported problems on the five EQ-5D health dimensions. A numerical value can be attached to each EQ-5D health state to reflect how good or bad a health state is according to the preferences of the general population of a country/region. The five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression).
NRS Numeric rating scale back pain and pain to the lower limbs | 12 months
  From the Norwegian quality register for spinal surgery. 0-10 pain scale for backpain and pain in the lower limbs. 0 represent no pain and 10 the worst pain ever.
Satisfaction og treatment and result on a 7 point likert scale | 12 months
  From the Norwegian quality register for spinal surgery.
  1. Complete recovered
  2. A lot better
  3. A bit better
  4. No change
  5. A bit worse
  6. A lot worse
  7. Worse than ever

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M. Röhrl, PhD, Study Director — Oslo University Hospital
Locations (1):
- Ullevål University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Axelsson P, Karlsson BS. Intervertebral mobility in the progressive degenerative process. A radiostereometric analysis. Eur Spine J. 2004 Oct;13(6):567-72. doi: 10.1007/s00586-004-0713-5. Epub 2004 May 19. PMID 15150701
- [Background] Fayyazi AH, Ordway NR, Park SA, Fredrickson BE, Yonemura K, Yuan HA. Radiostereometric analysis of postoperative motion after application of dynesys dynamic posterior stabilization system for treatment of degenerative spondylolisthesis. J Spinal Disord Tech. 2010 Jun;23(4):236-41. doi: 10.1097/BSD.0b013e3181a4bb0b. PMID 20072031
- [Background] Nabhan A, Al-Yhary A, Ishak B, Steudel WI, Kollmar O, Steimer O. Analysis of spinal kinematics following implantation of lumbar spine disc prostheses versus fusion: radiological study. J Long Term Eff Med Implants. 2007;17(3):207-16. doi: 10.1615/jlongtermeffmedimplants.v17.i3.40. PMID 19023945
- [Background] Sturesson B, Uden A, Vleeming A. A radiostereometric analysis of the movements of the sacroiliac joints in the reciprocal straddle position. Spine (Phila Pa 1976). 2000 Jan 15;25(2):214-7. doi: 10.1097/00007632-200001150-00012. PMID 10685486
- [Background] Sturesson B, Uden A, Vleeming A. A radiostereometric analysis of movements of the sacroiliac joints during the standing hip flexion test. Spine (Phila Pa 1976). 2000 Feb 1;25(3):364-8. doi: 10.1097/00007632-200002010-00018. PMID 10703111
- [Background] Zoega B, Karrholm J, Lind B. Plate fixation adds stability to two-level anterior fusion in the cervical spine: a randomized study using radiostereometry. Eur Spine J. 1998;7(4):302-7. doi: 10.1007/s005860050079. PMID 9765038
- [Background] Broden C, Olivecrona H, Maguire GQ Jr, Noz ME, Zeleznik MP, Skoldenberg O. Accuracy and Precision of Three-Dimensional Low Dose CT Compared to Standard RSA in Acetabular Cups: An Experimental Study. Biomed Res Int. 2016;2016:5909741. doi: 10.1155/2016/5909741. Epub 2016 Jul 10. PMID 27478832
- [Background] Broden C, Sandberg O, Skoldenberg O, Stigbrand H, Hanni M, Giles JW, Emery R, Lazarinis S, Nystrom A, Olivecrona H. Low-dose CT-based implant motion analysis is a precise tool for early migration measurements of hip cups: a clinical study of 24 patients. Acta Orthop. 2020 Jun;91(3):260-265. doi: 10.1080/17453674.2020.1725345. Epub 2020 Feb 14. PMID 32056507
- [Background] Nagamoto Y, Iwasaki M, Sakaura H, Sugiura T, Fujimori T, Matsuo Y, Kashii M, Murase T, Yoshikawa H, Sugamoto K. Sacroiliac joint motion in patients with degenerative lumbar spine disorders. J Neurosurg Spine. 2015 Aug;23(2):209-16. doi: 10.3171/2014.12.SPINE14590. Epub 2015 May 15. PMID 25978076
- [Background] Forsth P, Svedmark P, Noz ME, Maguire GQ Jr, Zeleznik MP, Sanden B. Motion Analysis in Lumbar Spinal Stenosis With Degenerative Spondylolisthesis: A Feasibility Study of the 3DCT Technique Comparing Laminectomy Versus Bilateral Laminotomy. Clin Spine Surg. 2018 Oct;31(8):E397-E402. doi: 10.1097/BSD.0000000000000677. PMID 29939843
- [Background] Svedmark P, Berg S, Noz ME, Maguire GQ Jr, Zeleznik MP, Weidenhielm L, Nemeth G, Olivecrona H. A New CT Method for Assessing 3D Movements in Lumbar Facet Joints and Vertebrae in Patients before and after TDR. Biomed Res Int. 2015;2015:260703. doi: 10.1155/2015/260703. Epub 2015 Oct 26. PMID 26587533
- [Background] Svedmark P, Tullberg T, Noz ME, Maguire GQ Jr, Zeleznik MP, Weidenhielm L, Nemeth G, Olivecrona H. Three-dimensional movements of the lumbar spine facet joints and segmental movements: in vivo examinations of normal subjects with a new non-invasive method. Eur Spine J. 2012 Apr;21(4):599-605. doi: 10.1007/s00586-011-1988-y. Epub 2011 Sep 1. PMID 21881866
- [Background] Eriksson T, Maguire GQ Jr, Noz ME, Zeleznik MP, Olivecrona H, Shalabi A, Hanni M. Are low-dose CT scans a satisfactory substitute for stereoradiographs for migration studies? A preclinical test of low-dose CT scanning protocols and their application in a pilot patient. Acta Radiol. 2019 Dec;60(12):1643-1652. doi: 10.1177/0284185119844166. Epub 2019 May 1. No abstract available. PMID 31042065
- [Background] Kibsgard TJ, Rohrl SM, Roise O, Sturesson B, Stuge B. Movement of the sacroiliac joint during the Active Straight Leg Raise test in patients with long-lasting severe sacroiliac joint pain. Clin Biomech (Bristol). 2017 Aug;47:40-45. doi: 10.1016/j.clinbiomech.2017.05.014. Epub 2017 May 29. PMID 28582642
- [Background] Kibsgard TJ, Roise O, Stuge B, Rohrl SM. Precision and accuracy measurement of radiostereometric analysis applied to movement of the sacroiliac joint. Clin Orthop Relat Res. 2012 Nov;470(11):3187-94. doi: 10.1007/s11999-012-2413-5. Epub 2012 Jun 14. PMID 22695864